CLINICAL TRIAL: NCT04562883
Title: Effect of Single vs. Group CAPA-IVM Culture of Human Cumulus-oocyte Complexes From Small Antral Follicles in a SIBLING Oocyte Study Design
Brief Title: Single vs. Group CAPA-IVM Culture of Cumulus-oocyte Complexes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mỹ Đức Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13/20/DD-BVMD
Record Dates: First submitted 2020-09-05; First posted 2020-09-24 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: IVF; PCOS; IVM
Keywords: CAPA-IVM; Single culture; Group culture
MeSH Terms: interventions — Culture Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single Culture (Experimental): Transfer the COCs cultured individually in Capacitation medium to the individual washing droplets from the "washing dish" containing "Maturation Medium" and wash them thoroughly. Then transfer COCs one by one to the "Culture dish" with "Maturation Medium".
  Interventions: Other: The way of Cumulus-oocyte complexes (COC) culture
- Group Culture (Experimental): Transfer half of the COCs (5-10 at a time) from the Capacitation culture dish to the "washing dish" containing "Maturation Medium (Group Culture)" by using an Eppendorf micropipette and wash them thoroughly (load pipette tips with 5µl, max. 10µl). Then transfer COCs to the "IVM dish" with "Maturation Medium (Group Culture)".
  Interventions: Other: The way of Cumulus-oocyte complexes (COC) culture

INTERVENTIONS:
Other: The way of Cumulus-oocyte complexes (COC) culture — Cumulus-oocyte complexes (COC) will be cultured in CAPA-IVM standard conditions: 24 hrs capacitation followed by 30h maturation. The first group will be culture in pools (group culture). The second group will be culture individually in 20µl droplets.

SUMMARY:
Oocyte in vitro maturation (IVM) is a minimal-stimulation ART with reduced hormone-related side effects and risks for the patients. However, the approach is not widely used because of an efficiency gap compared to conventional ART. In order to further optimize and adapt the CAPA-IVM system in the IVM clinic, this pilot study aims to check the feasibility of applying a single COC CAPA-IVM strategy versus the group COC culture CAPA-IVM

DETAILED DESCRIPTION:
Oocyte in vitro maturation (IVM) is a minimal-stimulation ART with reduced hormone-related side effects and risks for the patients. However, the approach is not widely used because of an efficiency gap compared to conventional ART.

Oocytes retrieved for IVM procedures derive from a heterogeneous pool with variable cellular and molecular characteristics that indicate its immature status. Thus, in vitro systems that permit and enhance acquisition and synchronization of meiotic competence (ability to resume meiosis in response to an ovulatory stimulus) and developmental competence (ability to be fertilized and support early embryo development) before the meiotic trigger are crucial for the optimization of human IVM systems.

A novel two-step IVM culture system (named CAPA-IVM) involving a pre-maturation culture with C-type natriuretic peptide (CNP) and a maturation step in presence of Amphiregulin (AREG), both more physiological compounds improving oocyte competence, have been introduced in previous clinical studies. So far these pilot studies proved to increase the rates of oocyte maturation, good quality embryos on day 3, good quality blastocyst, and as a result a higher embryo yield. CAPA-IVM blastocysts have shown similar rates of methylation and gene expression at gDMRs compared to COS embryos; and the expression of ma-jor epigenetic regulators was similar between both groups. Furthermore, an improvement in pregnancy rates strengthens the clinical relevance of the use of CAPA-IVM strategy.

In order to further optimize and adapt the CAPA-IVM system in the IVM clinic, this pilot study aims to check the feasibility of applying a single COC CAPA-IVM strategy versus the group COC culture CAPA-IVM. A single COC culture would permit to perform a non-invasive molecular analysis per matured oocyte, in order to identify quality genes ex-pressed in cumulus cells post-IVM (cumulus biomarkers), which could be subsequently used to identify the embryo(s) with highest potential of implantation.

ELIGIBILITY:
Inclusion Criteria:

* Having polycystic ovarian morphology: at least 25 follicles (2-9 mm) throughout the whole ovary and/or increased ovarian volume (>10ml) (it is sufficient that 1 ovary fits these criteria)
* No major uterine or ovarian abnormalities
* Having at least 15 follicles on the OPU day
* Patients consent to participate in the study

Exclusion Criteria:

* High (>grade 2) grade endometriosis
* Cases with extremely poor sperm (serve OAT: density <1 million, mobility <10% and sperm from testicular surgery)

Ages: 18 Years to 37 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2021-10-24 (Actual)

PRIMARY OUTCOMES:
Number of good quality embryos | At least 3 days after intra-cytoplasmic sperm injection
  Number of good quality Day 3 embryos obtained

SECONDARY OUTCOMES:
Maturation rate | Two days after oocytes pick-up
  Percentage of mature oocytes by 2 types of COC culture
Fertilization rate | 16-18 hours after intra-cytoplasmic sperm injection
  Percentage of fertilized oocytes by 2 types of COC culture
Cleavage rate | At least 3 days after intra-cytoplasmic sperm injection
  Percentage of day-3 embryos over fertilized oocytes by 2 types of COC culture
Expansion rate | After at least 30 hours of maturation culture
  Percentage of cumulus-oocyte complexes expanded after culture by 2 types of COC culture
The relative expression ratio ( R ) of human cumulus cell genes | cumulus cells will be collected after at least 30 hours of maturation culture, storaged at -80oC until RNA purification
  Cumulus cells will be collected, cDNA synthesis after mRNA purification, relative quantification PCR for detecting gene expression
Positive pregnancy test | at 2 weeks after the embryo placement after the completion of the first transfer
  Serum human chorionic gonadotropin level greater than 25 mIU/mL
Clinical pregnancy | 5 weeks after embryo placement after the completion of the first transfer
  at least one gestational sac on ultrasound at 7 weeks' gestation with the detection of heart beat activity
Ongoing pregnancy | At 12 weeks' gestation
  Ongoing pregnancy is defined as pregnancy with detectable heart rate at 12 weeks' gestation or beyond, after the completion of the first transfer
Implantation rate | 3 weeks after embryo transferred after the completion of the first transfer
  as the number of gestational sacs per number of embryos transferred
Multiple pregnancy | 5 weeks after embryo placement after the completion of the first transfer
  Defined as presence of more than one sac at early pregnancy ultrasound (6-8 weeks gestation)
Multiple delivery | At 24 weeks' gestation
  Birth of more than one baby beyond 24 weeks
Miscarriage | at 24 weeks of gestation after the completion of the first transfer
  pregnancy loss at < 24 weeks
Live birth | At 24 weeks of gestation
  defined as at least one newborn after 24 weeks of gestation and exhibiting any sign of life; twins were counted as a single birth

CONTACTS AND LOCATIONS:
Overall Officials: Tuong M Ho, MD, MCE, Principal Investigator — Hope Research Center
Locations (1):
- My Duc Hospital, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sanchez F, Le AH, Ho VNA, Romero S, Van Ranst H, De Vos M, Gilchrist RB, Ho TM, Vuong LN, Smitz J. Biphasic in vitro maturation (CAPA-IVM) specifically improves the developmental capacity of oocytes from small antral follicles. J Assist Reprod Genet. 2019 Oct;36(10):2135-2144. doi: 10.1007/s10815-019-01551-5. Epub 2019 Aug 9. PMID 31399916
- [Background] Vuong LN, Le AH, Ho VNA, Pham TD, Sanchez F, Romero S, De Vos M, Ho TM, Gilchrist RB, Smitz J. Live births after oocyte in vitro maturation with a prematuration step in women with polycystic ovary syndrome. J Assist Reprod Genet. 2020 Feb;37(2):347-357. doi: 10.1007/s10815-019-01677-6. Epub 2020 Jan 4. PMID 31902102
- [Background] Sanchez F, Romero S, De Vos M, Verheyen G, Smitz J. Human cumulus-enclosed germinal vesicle oocytes from early antral follicles reveal heterogeneous cellular and molecular features associated with in vitro maturation capacity. Hum Reprod. 2015 Jun;30(6):1396-409. doi: 10.1093/humrep/dev083. Epub 2015 Apr 22. PMID 25904637
- [Background] Saenz-de-Juano MD, Ivanova E, Billooye K, Herta AC, Smitz J, Kelsey G, Anckaert E. Genome-wide assessment of DNA methylation in mouse oocytes reveals effects associated with in vitro growth, superovulation, and sexual maturity. Clin Epigenetics. 2019 Dec 19;11(1):197. doi: 10.1186/s13148-019-0794-y. PMID 31856890
- [Result] Sanchez F, Lolicato F, Romero S, De Vos M, Van Ranst H, Verheyen G, Anckaert E, Smitz JEJ. An improved IVM method for cumulus-oocyte complexes from small follicles in polycystic ovary syndrome patients enhances oocyte competence and embryo yield. Hum Reprod. 2017 Oct 1;32(10):2056-2068. doi: 10.1093/humrep/dex262. PMID 28938744